CLINICAL TRIAL: NCT00508495
Title: Single-Dose Comparison of the Analgesic Efficacy, Safety and Tolerability of Two Paracetamol 1%-Containing Solutions and Placebo in a Post-Surgical Total Hip Replacement Model
Brief Title: Analgesic Efficacy, Safety and Tolerability of Two Paracetamol-Containing Solutions in Post-Surgical Hip Replacement Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: MDS Pharma Services (Industry)
Responsible Party: Keyvan Tadjalli Mehr, MD, MSc/Medical Director, Baxter Deutschland GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-01270-A016; EudraCT 2006-004075-36
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Pain, Postoperative
Keywords: pain, postoperative; replacement, total hip; total hip replacement; arthroplasty, replacement, hip
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Solutions; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test drug (Experimental)
  Interventions: Drug: Paracetamol 1% solution
- Reference drug (Active Comparator)
  Interventions: Drug: Paracetamol (acetaminophen)
- Placebo (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride solution

INTERVENTIONS:
Drug: Paracetamol (acetaminophen) — Four 100 mL, 15 min IV infusions at six hour intervals
  Other Names: Perfalgan
  Arms: Reference drug
Drug: Paracetamol 1% solution — Four 100 mL, 15 min IV infusions at six hour intervals
  Arms: Test drug
Drug: 0.9% sodium chloride solution — Four 100 mL, 15 min IV infusions at six hour intervals
  Other Names: Normal saline solution
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the therapeutic efficacy, safety and local tolerability of two different paracetamol-containing solutions in postoperative total hip replacement. They will be compared to placebo (a dummy treatment which contains no active ingredient).

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II or III and scheduled for elective total hip replacement, using a standard approach and a cemented implant.
* Moderate or severe pain within 4 hours after stopping the PCA in the morning of the first post-operative day.

Exclusion Criteria:

* Another acute or chronic painful physical condition
* Use of any other analgesics (within 24 hours), sedatives, or narcotic drugs as well as microsomal enzyme inducers
* Inability to use and understand Visual Analog Scale and Verbal Rating Score

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Amount of PCA-administered morphine consumed during first six hours of study drug treatment | 6 hours from first (of four) study drug doses

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Tadjalli Mehr, MD, MSc, Study Director — Baxter Deutschland GmbH
Locations (8):
- Hungary (8):
  - Réthy Pál Kórház-Rendelőintézet, Békéscsaba
  - Semmelweis Egyetem Ortopédiai Klinika, Budapest
  - Esztergom Város Önkormányzat Vaszary Kolos Kórháza, Esztergom
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Bács-Kiskun Megyei Önkormányzat Kórháza, Kecskemét
  - SZTE ÁOK Ortopédiai Klinika, Szeged
  - Tolna Megyei Önkormányzat Balassa János Kórháza, Szekszárd
  - Fejér Megyei Szent György Kórház, Székesfehérvár